CLINICAL TRIAL: NCT03780231
Title: Effect of Intense Sport Practice in Athletes With Non-ischemic Scar
Acronym: EISCAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3026_EISCAR
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Athletes With Isolated Non-ischemic LGE With no Underlying "Labelled" Cardiomyopathy
Keywords: Athletes; Late gadolinium enhancement; fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-ischemic scar — non-ischemic LGE with no underlying "labelled" cardiomyopathy is detected on CMR

SUMMARY:
The prognostic relevance of isolated non-ischemic LGE (i.e. with no underlying "labelled" cardiomyopathy) is unclear, and current guidelines to not state on the clearance of athlete with this type of findings as regards to competitive or intense sport practice.

The principal objective of the study is to evaluate during a five-years follow up, the clinical outcome of athletes with this kind of findings. The secondary objective is the determination of prognostic factors. The management and follow-up of the athletes will be let at the appraisal of each center.

DETAILED DESCRIPTION:
The presence of a scar, assessed by late gadolinium enhancement (LGE) on cardiac resonance imaging (CMR), is associated with a poor prognosis in patients with ischemic heart disease or cardiomyopathy. But the prognostic relevance of isolated non-ischemic LGE (i.e. with no underlying "labelled" cardiomyopathy) is unclear, and current guidelines do not state on the clearance of athlete with this type of findings as regards to competitive or intense sport practice.

The objective of the study is to evaluate the clinical outcome of athletes with isolated non-ischemic LGE with no underlying "labelled" cardiomyopathy during a five-years follow-up. The secondary objective is the determination of prognostic factors based on the baseline inclusion data: indication of CMR (i.e. symptoms, abnormal ECG, presence and morphology of arrhythmias, abnormal echocardiography); localization and amount of LGE, left and right ventricular geometry and function, characteristics of sport practice (amount, type, competition).

The management of the athletes will be let at the appraisal of each centre, as regards to the initial assessment, the follow-up and the medical clearance for competitive sports participation. Nevertheless, due to the absence of consensus, we propose that the patient should at least undergo clinical examination, ECG, echocardiography, cardiopulmonary exercise test (CPET) and holter ECG each year. A CMR should be performed at one and five years.

ELIGIBILITY:
Inclusion Criteria:

* Any athlete, aged of more than 15 years, symptomatic or not,
* in whom non-ischemic LGE with no underlying "labelled" cardiomyopathy is detected on CMR. Scare of an acute myocarditis will also be included.

Athletes will be defined by a practice of ≥4 hours/week of sport activity and/or competitive sport activity at the time of the assessment which triggered the realization of the 1st CMR.

Exclusion Criteria:

* Athletes with any unequivocal cardiac disease that might explain the LGE (i.e. hypertrophic cardiomyopathy, ischemic cardiac disease). In case of borderline or doubtful diagnosis the athlete can still be included (for example an athlete with a dilated LV and borderline function, or with borderline wall thickness).
* Patients who refuse their participation in the study.
* Patients under legal protection or deprived of their liberty.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any athlete, aged of more than 15 years, symptomatic or not, in whom non-ischemic LGE with no underlying "labelled" cardiomyopathy is detected on CMR.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-10-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a major cardiac event | five years after inclusion
  During a follow-up of 5 years, occurrence of a major cardiac event defined by either: death, death of cardiovascular cause; hospitalization for cardiac event; any major arrhythmic event defined by arrhythmic cardiac arrest, sustained ventricular tachycard

SECONDARY OUTCOMES:
Morphological end-point | five years after inclusion
  Alteration of left ventricular (LV) function defined by a decrease in LVEF as compared to the initial evaluation (≥10%, or occurrence of a new wall motion abnormality assessed the same imaging technic, i.e. echocardiography or CMR)
Functional end-point | five years after inclusion
  alteration of exercise capacity, defined by a reduction ≥10% of peak VO2, not explained by training changes
Arrhythmic end-point | five years after inclusion
  Occurrence of a non-sustained VT (NSVT), defined as a tachycardia originating in the ventricle >100 beats/min and lasting ≥3 beats but less than 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic FC SCHNELL, MD, Study Director — Rennes University Hospital
Locations (6):
- Baker IDI Heart and Diabetes Institute, Melbourne, Australia
- University Hospital Gasthuisberg, Leuven, Belgium
- CHU de Rennes, Rennes, France
- Saarland University, Saarbrücken, Germany
- Hospital Center of Luxembourg, Luxembourg, Luxembourg
- St. George's University of London, London, United Kingdom